CLINICAL TRIAL: NCT06512285
Title: Identification of Oxygen Desaturation in Patients Admitted Following Adenotonsillectomy'
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Adam Adler MD, MS, FAAP, Associate Professor of Anesthesiology, Baylor College of Medicine
Other Study IDs: H-53724
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adenotonsillectomy patients: Patients having undergone adenotonsillectomy at Texas Children's Hospital admitted for overnight observation based on our institutional protocol will be enrolled. A Wrist OX 3150 (Nonin Medical) will be placed in PACU with saturations recorded until the following morning after the surgery. The patient will undergo pulse oximetry monitoring separately based on the hospital protocol that will be used to guide care. Data from the Wrist Ox will not be avail to the treatment team and will only be analyzed for research purposes.
  Interventions: Diagnostic Test: Continuous Pulse Oximetry

INTERVENTIONS:
Diagnostic Test: Continuous Pulse Oximetry — The patient will wear a continuous pulse oximeter after their adenotonsillectomy surgery until the following morning. This will record continuous pulse oximetry data to allow for analysis of any desaturations in the first night following the surgery. This study is observational only and this data will not be used to impact any treatment

SUMMARY:
Sleep apnea has become exceedingly recognized in children. The primary treatment for sleep apnea in children is surgery in the form of adenotonsillectomy. The majority of children that undergo adenotonsillectomy are discharged following their immediate recovery in the post anesthesia care unit.

DETAILED DESCRIPTION:
Based on national and international consensus statements, institutional practice has developed at Texas Children's Hospital as to which patients require overnight observation following adenotonsillectomy for continuous pulse oximeter monitoring to assess for desaturation events. There is insufficient evidence to suggest which patients need to stay for pulse oximeter monitoring which has led to many patients being admitted unnecessarily. Therefore, the aim of this study is to capture data prospectively on pulse oximetry in children admitted overnight following adenotonsillectomy to identify risk factors for post operative oxygen desaturation.

ELIGIBILITY:
Inclusion Criteria:

* Adenotonsillectomy surgery
* Patient meeting institutional guidelines for postoperative admission (e.g, admitted following surgery from recovery room).

Exclusion Criteria:

* Parental refusal
* Airway Surgery in addition to adenotonsillectomy
* Patient psychological limitations, precluding wearing device (e.g. autism).
* Patient not meeting institutional guidelines for postoperative admission (e.g, discharged following surgery from recovery room).

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing adenotonsilectomy at Texas Children's Hospital Main campus that meet institutional requirements for post-operative admission for continuous pulse oximetry monitoring
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2024-07-25 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Continuous pulse oximetry following adenotonsillectomy | 1 day
  Use of a continuous capture pulse oximeter to identify oxygen desaturations postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: adam adler, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Childrens Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified data will be shared on reasonable written request to the PI. in accordance with institutional policies